CLINICAL TRIAL: NCT00254904
Title: International, Randomized, Open-Label, Phase 3 Trial of Gemcitabine/Cisplatin Plus PF-3512676 Versus Gemcitabine/Cisplatin Alone as First-Line Treatment of Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Randomized Trial of Gemcitabine/Cisplatin + PF-3512676 vs Gemcitabine/Cisplatin Alone in Patients With Advanced NSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Termination Reason in Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8501002
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: advanced carcinoma, non-small cell lung, Phase III, Gemcitabine, Gemzar, Cisplatin, Platinol, PF-3512676, immunotherapy, immune modulator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Standard of Care chemotherapy plus experimental intervention (PF-3512676)
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: PF-3512676
- B (Active Comparator): Standard of Care chemotherapy
  Interventions: Drug: Cisplatin; Drug: Gemcitabine + Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 75 mg/m2 intravenously on day 1 of each 21 day cycle x 6 cycles
  Other Names: Platinol-AQ
  Arms: A
Drug: Gemcitabine — Gemcitabine 1250 mg/m2 intravenously on days 1 and 8 of each 21 cycle x 6 cycles
  Other Names: Gemzar
  Arms: A
Drug: PF-3512676 — PF-3512676 0.2 mg/kg subcutaneously days 8 and 15 x 6 cycles and then weekly until disease progression or unacceptable toxicity
  Arms: A
Drug: Cisplatin — Cisplatin 75 mg/m2 intravenously on day 1 of each 21 day cycle x 6 cycles
  Other Names: Platinol-AQ
  Arms: B
Drug: Gemcitabine + Cisplatin — Gemcitabine 1250 mg/m2 intravenously on days 1 and 8 of each 21 cycle x 6 cycles
  Other Names: Gemzar
  Arms: B

SUMMARY:
To assess the efficacy and safety of PF-3512676 administered in combination with gemcitabine/cisplatin chemotherapy as first-line treatment in patients with locally advanced or metastatic Non-Small-Cell Lung Cancer (NSCLC) and to compare it to the efficacy and safety of gemcitabine/cisplatin alone.

DETAILED DESCRIPTION:
PF-3512676 dosing was stopped 20 June 2007 in response to DSMC recommendation to close the trial, citing lack of efficacy concerns as the primary reason with a safety issue (thrombocytopenia) also contributing to the decision. Subjects were allowed to complete standard of care treatment/survival follow-up. Data collection was completed on 25 June 2008.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-Small-Cell Lung Cancer (NSCLC) stage IIIB with pleural effusion or stage IV
* No prior systemic treatment for Non-Small-Cell Lung Cancer (NSCLC) with chemotherapy, immunotherapy, biologic response modifiers or other investigational drugs
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1

Exclusion Criteria:

* Small cell or carcinoid lung cancer
* Known Central Nervous System (CNS) metastasis
* Pre-existing auto-immune or antibody mediated diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 656 Events

SECONDARY OUTCOMES:
Patient Reported Outcomes | End of treatment
Overall Safety Profile | 28 days post PF03512676 dosing
Progression Free Survival | Time of primary endpoint
Time to Tumor Progression | Time of progressive disease
Overall Objective Response | End of treatment
Duration of Response | Time of progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (103):
- United States (7):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Bakersfield, California
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Spokane, Washington
- Pfizer Investigational Site, Innsbruck, Austria
- Belgium (6):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Charleroi
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Jette
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
- Brazil (3):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Jaú, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (6):
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Lévis, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- China (4):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Dalian, Liaoning
  - Pfizer Investigational Site, Beijing
- Czechia (3):
  - Pfizer Investigational Site, Prague, CZ
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Prague
- Germany (6):
  - Pfizer Investigational Site, Bielefeld
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Löwenstein
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Tübingen
- Hong Kong (2):
  - Pfizer Investigational Site, Kowloon
  - Pfizer Investigational Site, Shatin
- Hungary (5):
  - Pfizer Investigational Site, Zalaegerszeg, Külsőkórház-Pózva
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Deszk
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Pécs
- India (6):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, New Delhi, New Delhi
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh
- Israel (2):
  - Pfizer Investigational Site, Beersheba
  - Pfizer Investigational Site, Kfar Saba
- Italy (5):
  - Pfizer Investigational Site, Forlì
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, S.Andrea Delle Fratte (PG)
- Netherlands (5):
  - Pfizer Investigational Site, Amsterdam, North Holland
  - Pfizer Investigational Site, Zaandam, North Holland
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Harderwijk
  - Pfizer Investigational Site, Nijmegen
- Poland (6):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Otwock
  - Pfizer Investigational Site, Szczecin-Zdunowo
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wodzislaw Sl.
- Portugal (3):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Slovakia (4):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Kvetnica Pri Poprade
  - Pfizer Investigational Site, Nitra-Zobor
- South Africa (3):
  - Pfizer Investigational Site, Port Elizabeth, Eastern Cape
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Port Elizabeth
- South Korea (2):
  - Pfizer Investigational Site, Gyeonggi-do
  - Pfizer Investigational Site, Seoul
- Spain (7):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Castellon, Castellon
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Jaén, Jaen
  - Pfizer Investigational Site, Barakaldo, Vizcaya
- Taiwan (3):
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei
- Turkey (Türkiye) (3):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Bornova / Izmir
  - Pfizer Investigational Site, Istanbul / Ceraahpasa
- United Kingdom (10):
  - Pfizer Investigational Site, Bristol, Avon
  - Pfizer Investigational Site, Southampton, Hampshire
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Wolverhampton

REFERENCES:
- [Derived] Roeland EJ, Fintelmann FJ, Yang R, Tarasenko L, Bonomi PD. Evaluation of Weight Gain and Overall Survival of Men Versus Women With Advanced Non-Small Cell Lung Cancer. J Cachexia Sarcopenia Muscle. 2025 Dec;16(6):e70131. doi: 10.1002/jcsm.70131. PMID 41332393
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8501002&StudyName=Randomized%20trial%20of%20gemcitabine/cisplatin%20+%20PF-3512676%20vs%20gemcitabine/cisplatin%20alone%20in%20patients%20with%20advanced%20NSCLC%20